CLINICAL TRIAL: NCT06866600
Title: Study on the Safety and Efficacy of Human IPSC-Derived Cardiomyocytes in the Treatment of End-Stage Heart Failure
Brief Title: IPSC-CMs Combined with LVAD or CABG for the Treatment of Heart Failure
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Help Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYF, WLS
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure; Heart Failure At NYHA Stage III or IV
Keywords: LVAD; CABG; iPSC-CMs
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (Sham Comparator): CABG combined with saline or LVAD combined with saline
  Interventions: Other: CABG/LVAD+Saline
- Low Dose Group (Experimental): CABG combined with 0.5×10^8 iPSC-CMs
  Interventions: Biological: low dose CABG+iPSC-CMs
- High dose group (Experimental): CABG combined with 1.5×10^8 iPSC-CMs or LVAD combined with 1.5×10^8 iPSC-CMs
  Interventions: Biological: High dose CABG/LVAD+iPSC-CMs

INTERVENTIONS:
Biological: low dose CABG+iPSC-CMs — CABG+0.5×10^8 iPSC-CMs
  Arms: Low Dose Group
Biological: High dose CABG/LVAD+iPSC-CMs — CABG+1.5×10^8 iPSC-CMs or LVAD+1.5×10^8 iPSC-CMs
  Arms: High dose group
Other: CABG/LVAD+Saline — CABG/LVAD+Saline
  Arms: Control group

SUMMARY:
This clinical trial investigates the safety, feasibility, and therapeutic potential of a combined approach using HiCM-188 cardiomyocyte injection delivered intramyocardially alongside either LVAD implantation or CABG surgery in patients with advanced ischemic heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 35-75 years (inclusive) at the time of signing the informed consent form.
* Capable of understanding the informed consent form, voluntarily agreeing to participate in the trial, and signing the informed consent form.
* Diagnosed with end-stage heart failure.
* Receiving optimized medical therapy for heart failure, with New York Heart Association (NYHA) functional class III-IV.
* Echocardiography demonstrating regional hypokinesia or akinesia of the ventricular wall.
* Cardiac magnetic resonance imaging (MRI) confirming left ventricular ejection fraction (LVEF) ≤35%.
* Myocardial perfusion-metabolism imaging with radionuclide indicating infarcted myocardium in the left anterior descending (LAD) artery territory.
* Meets criteria for coronary artery bypass grafting (CABG) under cardiopulmonary bypass during screening and requires CABG surgery.
* For patients enrolled in the LVAD implantation group, the following additional criteria must be met:

  1. Definitive indication for LVAD implantation due to end-stage heart failure.
  2. Anticipated significant improvement in hemodynamic stability post-LVAD implantation, with potential for further cardiac functional improvement via myocardial cell injection.
  3. Absence of significant contraindications for LVAD surgery.

Exclusion Criteria:

* History of pacemaker, implantable cardioverter-defibrillator (ICD), or cardiac resynchronization therapy (CRT).
* Severe valvular heart disease.
* Acute myocardial infarction or history of percutaneous coronary intervention (PCI) within 1 month prior to screening.
* Non-ischemic cardiomyopathy or acute viral myocarditis.
* Acute cerebrovascular event within 1 month prior to screening.
* History of malignancy within 5 years prior to screening.
* Autoimmune disease or chronic use of immunosuppressive agents.
* History of organ transplantation.
* Planned concurrent major surgery (excluding left ventricular aneurysm resection or left atrial appendage closure/resection).
* Malignant ventricular arrhythmia.
* Contraindications for CABG surgery.
* Positive serology for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or Treponema pallidum antibody.
* Inability to undergo cardiac MRI or PET/CT imaging.
* Contraindications to immunosuppressive therapy or inability to comply with the protocol-specified immunosuppressive regimen.
* Hypersensitivity to mycophenolate sodium, mycophenolic acid, mycophenolate mofetil, tacrolimus, macrolides, prednisone acetate/methylprednisolone, other corticosteroids, or basiliximab.
* Participation in another clinical trial within 3 months prior to screening.
* Pregnancy, lactation, or positive pregnancy test in female patients.
* Any other condition deemed by the investigator to render the patient unsuitable for trial participation.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
6-minute walk test | baseline, 1, 3, 6, 12 months post-operation
Major Adverse Cardiovascular Events | From enrollment to the end of study at 12 months
  The composite endpoint events occurring during the prescribed postoperative follow-up period included cardiac death, non-fatal myocardial infarction, non-fatal stroke, and emergency target vessel revascularization (e.g., PCI or CABG), which was expressed as the percentage of subjects experiencing at least one of these events (%).
Survival rate | From enrollment to the end of study at 12 months

SECONDARY OUTCOMES:
Left ventricular ejection fraction | baseline, 1, 3, 6, 12 months post-operation
  Improvement of left ventricular ejection fraction assessed by ECHO
Cardiac magnetic resonance detection index | baseline, 1, 3, 6, 12 months post-operation
  Myocardial infarction size and Myocardial fibrosis assessed by MRI
BNP | baseline, 1, 3, 6, 12 months post-operation
  BNP levels are measured by venous blood samples
SF-36 | baseline, 1, 3, 6, 12 months post-operation
  life quality assessed by SF-36 (The Short-Form-36 Health Survey). The SF-36 scale is a tool used to assess health-related quality of life, including eight dimensions: Physical Functioning (PF), Role-Physical (RP), Bodily Pain (BP), General Health (GH), Vitality (VT), Social Functioning (SF), Role-Emotional (RE), and Mental Health (MH). Each dimension has its unique scoring criteria, and the score range for each dimension is from 0 to 100 points. Higher scores indicate better health outcomes
KCCQ | baseline, 1, 3, 6, 12 months post-operation
  Kansas City Cardiomyopathy Questionnaire, KCCQ is designed to assess the health status and quality of life of patients with heart failure. The score range is from 0 to 100 and higher scores reflect better health status and quality of life.
Removal rate of LVAD | From enrollment to the end of study at 12 months
  Percentage of subjects who had their Left Ventricular Assist Device (LVAD) successfully removed after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yongfeng Shao, MD, PhD, Principal Investigator — Jiangsu Provincial People's Hospital (First Affiliated Hospital of Nanjing Medical University); Liansheng Wang, MD, PhD, Principal Investigator — Jiangsu Provincial People's Hospital (First Affiliated Hospital of Nanjing Medical University)
Locations (1):
- HelpThera, Nanjing, Jiangsu, China